CLINICAL TRIAL: NCT02669472
Title: Fresh to You: Multilevel Approaches in Low Income Housing to Increase F&V Intake
Acronym: LWVB
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: University of Connecticut (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Kim Gans, Principal Investigator/Adjunct Professor, Brown University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NCI; R01CA134903 (NIH)
Record Dates: First submitted 2016-01-19; First posted 2016-02-01 (Estimated); Last update posted 2016-02-01 (Estimated); Status verified 2016-01

CONDITIONS: Dietary Habits; Dietary Modification
MeSH Terms: conditions — Feeding Behavior | interventions — Milieu Therapy; Early Intervention, Educational; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- F&V Intervention (Experimental): Housing complexes randomized to the intervention arm received a multicomponent intervention comprised of a year-round, discount, mobile fresh fruit and vegetable market ('Fresh To You') that was paired with nutrition education interventions including educational newsletters, recipe cards, campaigns, taste-testings and videos in both English and Spanish.
  Interventions: Other: Environmental Intervention; Behavioral: Educational Intervention
- Control Intervention (Experimental): Housing complexes randomized to the comparison arm received a year-long intervention on physical activity and stress reduction including educational campaigns and materials in both English and Spanish.and a YMCA membership for those who joined the campaigns.
  Interventions: Behavioral: Control

INTERVENTIONS:
Other: Environmental Intervention — Intervention sites received regularly-scheduled, discount, fresh F&V markets for one year during the first two weeks of each month. The markets brought between 50-70 different produce items, including culturally desired ethnic produce. Markets at the senior and disabled housing complexes were held indoors as were markets at family housing complexes during inclement weather. In good weather, markets were held outside at the family complexes using a mobile retrofitted car trailer. The produce items were set up in racks on three sides of the trailer and shoppers entered through the rear door. FTY markets accepted cash, debit/credit cards and EBT cards (SNAP). Each market lasted two hours and the produce was sold at prices 15%-25% lower than local retail supermarket prices.
  Other Names: Fresh To You fruit and vegetable markets
  Arms: F&V Intervention
Behavioral: Educational Intervention — Each household in the housing site received a reusable shopping bag that contained a binder with: an overview page, sleeves to store 12 newsletters, three DVDs and 48 recipe cards. The 20-minute DVDs included cooking demonstrations, tips and testimonials. A two-page, full-color newsletter was delivered each household each month. It had information about a particular F&V in season as well as other tips and recipes. Two 6-week long educational and motivational campaigns were also offered: ''Just Add 2', and 'Color Your Plate'. Both campaigns included full-color campaign booklets, goal-setting activities, educational and motivational content, and F&V trackers with incentives/prizes for completing and turning in the trackers. All materials were provided in English and Spanish.
  Other Names: Nutrition education interventions
  Arms: F&V Intervention
Behavioral: Control — We contracted with the Greater Providence YMCA to bring to provide physical activity and stress reduction programming. Two, six-week campaigns followed the same format and timing of the intervention group campaigns. Campaigns participants received a free, 6-week membership to the YMCA. The 'Take 10!' campaign aimed to increase participants' daily physical activity by 10 minutes per day until they reached the goal of at least 30-60 minutes per day. The second campaign was 'Stress Less' aimed to help participants reduce the amount of stress that they experienced by including relaxation activity into their daily routine.
  Other Names: Physical Activity and Stress Reduction campaigns
  Arms: Control Intervention

SUMMARY:
Live Well, Viva Bien (LWVB) is an NCI-funded, cluster randomized controlled trial (RCT) that was conducted in 15 subsidized housing complexes to evaluate the efficacy of a multicomponent intervention comprised of a year-round, discount, mobile fresh F&V market -'Fresh To You' (FTY)- that was paired with a nutrition education component including included educational newsletters, campaigns, taste-testings and videos in both English and Spanish. The primary aim of the LWVB grant was to study the efficacy of FTY combined with a motivational/educational intervention to see if it increased F&V consumption compared to a Comparison intervention (attention placebo).

DETAILED DESCRIPTION:
'Live Well, Viva Bien' (LWVB) is a cluster randomized controlled trial in 15 subsidized housing complexes designed to evaluate the efficacy of a multicomponent intervention that includes discount, mobile fresh F&V markets--'Fresh To You'(FTY) markets-in conjunction with a nutrition education intervention. The primary aims of this study are to: 1) Conduct formative research with residents living in subsidized housing projects to inform the multi-level intervention and; 2) Implement a group randomized trial to study the efficacy of the FTY markets combined with the educational/motivational interventions at increasing F&V access, availability, and consumption compared to a Comparison intervention (attention placebo). Secondary aims are: 1) To include extensive implementation process evaluation to determine costs, reach, fidelity and dose and the relationship of these variables with evaluation outcomes; and to 2) Use a mediating variable framework to examine relationships among important psychosocial factors/determinants with changes in F&V consumption.

All study activities occurred at housing sites in Providence County, Rhode Island. Pre-intervention focus groups were conducted with housing complex residents (from non-study sites) to inform intervention development. A total of 15 subsidized housing complexes were recruited into the evaluation cohort. One smaller housing complex served as a pilot site for the intervention group and the remaining 14 demographically-matched sites were randomized into either the intervention or control group. Adult residents from each housing site were recruited for the evaluation cohort prior to randomization. The multicomponent intervention lasted one year and included baseline, 6 and 12 month follow-up surveys as well as extensive quantitative and qualitative process evaluation throughout the course of the study. All study protocols were approved by the Brown University Institutional Review Board.

The intervention sites received regularly-scheduled, discount, fresh F&V markets for one year. These FTY markets were not farmer's markets, but rather mobile markets selling both local and non-local produce on a year-round basis at prices at or below local supermarket prices. Intervention sites, markets received markets the first two weeks of each month. In addition, these Housing sites also received a motivational/educational intervention components over the course of the year including two campaigns (Just Add 2 and Color Your Plate), three, 20-minute DVDs, a two-page, full-color monthly newsletter , 48 Recipe cards, and cooking demonstrations at the housing sites.

The Comparison/Control Intervention sites received physical activity and stress reduction campaigns delivered by the Greater Providence YMCA.

Extensive process evaluation was conducted. Outcome measures included three different measures of F&V intake. Data on potential mediators and moderators was also conducted.

ELIGIBILITY:
Inclusion Criteria:

* Live in the Housing complex;
* Speak English or Spanish
* Ability to read study materials

Exclusion Criteria:

* Health issues that would not allow increases in fruit and vegetable intake

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1598 (Actual)
Dates: Start 2009-04; Primary Completion 2014-10 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change in Fruit and Vegetable Intake | Baseline, 6 and 12 months
  Measured by National Cancer Institute Eating at America's Table All Day Screener
Change in Fruit and Vegetable Intake | Baseline, 6 and 12 months
  Two-Item Cup F&V intake screener

SECONDARY OUTCOMES:
Change in fruit and vegetable behaviors | Baseline, 6 and 12 months
  F&V habits questions

IPD SHARING:
Plan to Share IPD: No
We will make aggregate data available to share.

REFERENCES:
- [Derived] Gans KM, Risica PM, Keita AD, Dionne L, Mello J, Stowers KC, Papandonatos G, Whittaker S, Gorham G. Multilevel approaches to increase fruit and vegetable intake in low-income housing communities: final results of the 'Live Well, Viva Bien' cluster-randomized trial. Int J Behav Nutr Phys Act. 2018 Aug 20;15(1):80. doi: 10.1186/s12966-018-0704-2. PMID 30126463
- [Derived] Gans KM, Gorham G, Risica PM, Dulin-Keita A, Dionne L, Gao T, Peters S, Principato L. A multi-level intervention in subsidized housing sites to increase fruit and vegetable access and intake: Rationale, design and methods of the 'Live Well, Viva Bien' cluster randomized trial. BMC Public Health. 2016 Jun 28;16:521. doi: 10.1186/s12889-016-3141-7. PMID 27353149